CLINICAL TRIAL: NCT03711201
Title: The Effects of the Preoperative Operating Room Environment Presentation on Preanesthetic Anxiety and Blood Pressure in Hypertensive Patients: A Prospective, Randomized Controlled Trial
Brief Title: Effects of Preoperative Operating Room Environment Presentation in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nureddin YUZKAT, Assist. prof., Yuzuncu Yil University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hypertensive patients
Record Dates: First submitted 2018-10-12; First posted 2018-10-18 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Hypertension; Anxiety; Blood Pressure
Keywords: Hypertensive patients; Introduction of operating room; Anxiety; Blood pressure
MeSH Terms: conditions — Hypertension; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group IORE (Active Comparator): This group will undergo the IORE procedure before surgery (operation). On the day of surgery, the patient will be brought to the operating room by the anesthesiologist. Hemodynamic data (blood pressure, pulse rate, respiratory rate, SpO2) will be measured at the service, preop unit and operating room. The anxiety level in the operating room will be measured by the ST-STAI scale.
  Interventions: Behavioral: Group IORE
- Group NoIORE (No Intervention): The patient's hemodynamic data will be measured in the evening service before surgery. The patient will be brought to the operating room by the anesthesiologist on the day of surgery and hemodynamic data (blood pressure, pulse rate, respiratory rate, SpO2) will be measured in the preop unit. The hemodynamic data and the ST-STAI scale will measure the anxiety level in the operating room.

INTERVENTIONS:
Behavioral: Group IORE — This group will undergo the IORE procedure before surgery (operation). On the day of surgery, the patient will be brought to the operating room by the anesthesiologist. Hemodynamic data (blood pressure, pulse rate, respiratory rate, SpO2) will be measured at the service, preop unit and operating room. The anxiety level in the operating room will be measured by the ST-STAI scale.
  Arms: Group IORE

SUMMARY:
The aim of this study was to investigate the effects of preoperative operating room environment introduction on preoperative hypertension and blood pressure in hypertensive patients.

DETAILED DESCRIPTION:
Procedure to be Applied:

In order to eliminate the other factors that cause essential HT, the patients' blood pressure due to HT should be controlled, the surgery will be planned as the first case in the morning and the patients will need 8 hours fasting period.

Patients' gender, age, height, weight values, ASA scores, body mass index (BMI) values will be recorded. Hemodynamic parameters (blood pressure, heart rate and SpO2 values) will be recorded in the services of the patients, in the preop unit and in the operation room. Hypertension requiring intervention or additional medication will be excluded from the study. A randomized number of patients will be included in the study according to the results of power analysis.

Introduction of the operating room environment (IORE): The procedure to be performed on the day of surgery will be simulated and accompanied by an anesthesiologist. The patient's hemodynamic data (blood pressure, pulse rate, respiratory rate, SpO2) will be measured at the time of operation, between 16: 00-18: 00 hours prior to the operation, and will be brought to the operating room with a service nurse. The hemodynamic data of the patient will be measured in the preop unit and the patient will be taken to the operating room with anesthesia doctor. Here, in addition to the patient's hemodynamic data, the instantaneous state anxiety scale (ST-STAI) will be completed and the patient will be left in service again. The procedure will be similar to the process that the patient will experience on the operation day.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* informed consent,
* essential hypertension was diagnosed,
* Between the ages of 40-80,
* American Society of Anesthesiologists (ASA) class II-III

Exclusion Criteria:

* drug allergy,
* with a history of malignant hyperthermia,
* uncontrolled hypertension,
* cancer and psychological problems,
* patients with cardiac and endocrine diseases
* emergency surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
anxiety | 1 day
  The patient's anxiety will be measured by instantaneous state anxiety scale (ST-STAI)

CONTACTS AND LOCATIONS:
Overall Officials: Nureddin Yüzkat, Study Chair — Yuzuncu Yil University Dursun Odabas Medical School Anesthesiology a nd Reanimation Department, Van, Turkey
Locations (1):
- Van yuzuncu Yıl University, Dursun Odabas Medical Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kakinuma A, Nagatani H, Otake H, Mizuno J, Nakata Y. The effects of short interactive animation video information on preanesthetic anxiety, knowledge, and interview time: a randomized controlled trial. Anesth Analg. 2011 Jun;112(6):1314-8. doi: 10.1213/ANE.0b013e31820f8c18. Epub 2011 Feb 23. PMID 21346166
- [Background] Shafer A, Fish MP, Gregg KM, Seavello J, Kosek P. Preoperative anxiety and fear: a comparison of assessments by patients and anesthesia and surgery residents. Anesth Analg. 1996 Dec;83(6):1285-91. doi: 10.1097/00000539-199612000-00027. PMID 8942601
- [Background] Paterniti S, Alperovitch A, Ducimetiere P, Dealberto MJ, Lepine JP, Bisserbe JC. Anxiety but not depression is associated with elevated blood pressure in a community group of French elderly. Psychosom Med. 1999 Jan-Feb;61(1):77-83. doi: 10.1097/00006842-199901000-00013. PMID 10024070